CLINICAL TRIAL: NCT03377075
Title: Study of the Choroidal and Retinal Thickness in Relation to Axial Length in Healthy Young Subjects With Swept-source Optical Coherence Tomography.
Brief Title: Study of the Choroidal and Retinal Thickness in Relation to Axial Length.
Acronym: CHORAL
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Miklos Schneider MD, PhD, Assistant Professor, Semmelweis University
Other Study IDs: CHORAL-1249
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy subjects
  Interventions: Device: AL measurement; Device: OCT

INTERVENTIONS:
Device: AL measurement — IOL Master 500 (Carl Zeiss AG, Germany)
Device: OCT — Choroidal and retinal thickness measurement (DRI OCT-1 Model Triton (plus), Topcon, Tokyo, Japan)

SUMMARY:
The aim of the study is the non-invasive morphological evaluation of the choroid and the retina in relation to the length of the eyeball in healthy, young man and women.

DETAILED DESCRIPTION:
The choroid is responsible for the oxygen supply of the outer retina, hence many diseases that affect the retina are originating from the choroid or at later stages influence the choroid as well. The functional efficiency of the choroid in a healthy subject is important. The thickness of the choroid is a marker for the extent of the vessels inside.

With optical coherence tomography (OCT) non-invasive and non-contact measurement of the choroidal and retinal thickness is possible. Swept-source OCT is one the latest developments of OCTs. Its increase wavelength allows deeper penetration than previous models and allows high resolution imaging.

OCTs are FDA approved machines, they are not considered experimental. The swept-source OCT machine (DRI OCT-1 Model Triton (plus), Topcon, Tokyo, Japan) used in the study is a CE marked commercially available medical device.

The goal of the study is to evaluate the choroidal and the retinal morphology in relation to the length of the eyeball (axial length - AL) in healthy, young adults.

There are several publications on this topic, most of them on asian populations.

In the study healthy, Caucasians in their twenties are recruited to minimize the aging effect on choroidal thickness.

Following informed consent, demographics are recorded, refraction is taken, axial length is measured with IOL Master 500 (Carl Zeiss AG, Germany) then OCT is performed.

Pupil dilation is not necessary. Images are stored digitally by abiding corresponding laws on personal data protection. Results are processed with statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, but less than 29 years of age
* Caucasian race
* Signed informed consent

Exclusion Criteria:

* Known epilepsy
* Inability to act
* Media opacity in the eye that would disturb imaging

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subject with no eye diseases.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Relation of choroidal thickness to axial length | Through study completion, 6 months
Relation of retinal thickness to axial length | Through study completion, 6 months

SECONDARY OUTCOMES:
Influence of age on results | Through study completion, 6 months
Influence of gender on results | Through study completion, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Schneider, Principal Investigator — Semmelweis University, Department of Ophthalmology
Locations (1):
- Semmelweis University, Department of Ophthalmology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No